CLINICAL TRIAL: NCT04213781
Title: Does Audiovisual Distraction Decrease the Use of Hypnotic Drugs During Oocyte Retrieval?
Brief Title: Interest of Audiovisual Distraction in the Management of Anxiety and Pain During Oocyte Retrieval
Acronym: Happy-Fiv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/02
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Fertilization in Vitro
Keywords: Oocyte retrieval; Sedation
MeSH Terms: interventions — Propofol; Sufentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Other): Sedation according to Dixon's up-and-down method.
  Interventions: Drug: Propofol; Drug: Sufentanil
- Audiovisual distraction (Experimental): Audiovisual distraction using HappyMed Video Glasses during procedure. Sedation according to Dixon's up-and-down method.
  Interventions: Device: HappyMed Video Glasses; Drug: Propofol; Drug: Sufentanil

INTERVENTIONS:
Device: HappyMed Video Glasses — HappyMed allows the immersion of patients in films, cartoons or concerts.
  Arms: Audiovisual distraction
Drug: Propofol — The dosage is modified according to the Dixon's up-and-down method (using 0.5 µg/ml as a step size). The first patient in each group will start at a dose 3 µg/ml propofol. If patient manifests discomfort then the next patient will receive an increment of 0.5 µg/ml propofol, if patient is comfortable, then the next patient received a decrement of 0.5 µg/ml propofol.
Drug: Sufentanil — 0.1 µg/kg

SUMMARY:
Oocyte retrieval procedure for in vitro fertilization is a source of anxiety for patients. Local anaesthesia or sedation are commonly used to manage many situations of anxiety, including the oocyte retrieval. However, this sedation should be as mild as possible in order to preserve oocytes.

HappyMed Video Glasses are a recent medical device that allows the immersion of patients in films, cartoons or concerts. By distracting patients, this technology can reduce anxiety, discomfort and ultimately pain associated with care.

This randomized monocentric trial compares audiovisual distraction versus usual care for the management of anxiety and pain related to oocyte retrieval.

Hypothesis of this study is that the audiovisual distraction carried out with the HappyMed Video Glasses reduces the use of sedative drugs during oocyte retrieval while ensuring a better comfort and a faster walking ability.

DETAILED DESCRIPTION:
Consent female patients between 18 and 43 years old scheduled for oocyte retrieval will be enrolled in this study and their anxiety level will be collected via a questionnaire.

After randomization, patients will either benefit from audiovisual distraction using HappyMed Video Glasses, (medical device with CE marking), or from the usual management during procedure. The anaesthesiologist will check that no anxiolytic or sedative drug was given 12 hours before anaesthesia. The patients will be stratified according to whether or not a previous intervention was performed. Anaesthesia will be started and maintained with administration of sufentanil (0.1 μg/kg) and propofol (using the Dixon's up-and-down method). The aim is a patient who spontaneously ventilates and does not react to gynaecological stimulation. Prevention of postoperative pain and nausea/vomiting will be carried out at the initiation of the surgical procedure. The effect of these drugs is longer than the intervention duration and will not influence the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing oocyte retrieval requiring a sedation associating sufentanil and propofol
* Contactable by phone the day after the procedure.
* Consent for participation
* Affiliation to the social security system

Exclusion Criteria:

* Corneal or conjunctival diseases in progress,
* Claustrophobia
* Patients under protection of the adults (guardianship, curators or safeguard of justice)
* Communication difficulties or neuropsychiatric disorder

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Target concentration of propofol administered during oocyte retrieval procedure to maintain the patient comfortable | Intraoperative period : from the start of anaesthesia to the end of the intervention
  An up and down method will define the CP 50 in each group.

SECONDARY OUTCOMES:
Side effects due to audiovisual distraction | 4 hours
  Onset of vertigo, nausea or headaches
Patient comfort during propofol injection | 30 minutes
  Comfort behavior scale : it incorporates three categories of behavior : Facial expression (0=relaxed ; 1= frowning ; 2=grimacing) ; Verbal response (0=none ; 1= moans ; 2=verbal protest) ; Arm movement (0=none ; 1=medium ; 2=strong). Each scored on a 0-2-point scale so that the total score ranges from 0 to 6.
Complications due to anaesthesia | up to 24 hours (from the start of anaesthesia to the patient's discharge of the recovery room)
  Occurence of desaturation event (SpO2< 92%), respiratory distress event (RR<10 breaths per minute) or bronchospasm.
Resumption of walking | 12 hours
  Duration between the end of the procedure and the standing position.
Health staff satisfaction | 2 hours
  Satisfaction VRS ranging from 0 to 4 (0=unsatisfied, 4=very satisfied).
Patient satisfaction | 4 hours
  Satisfaction VRS ranging from 0 to 4 (0=unsatisfied, 4=very satisfied).
Resuming activities of daily living | 24 hours
  Numeric scale from 0 to 10 (0=bedridden, 10=resuming total activities).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital FOCH, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No